CLINICAL TRIAL: NCT01322321
Title: A Randomized, Double-blind, Multiple-dose, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of ACZ885 in Patients With Newly Diagnosed Type-1 Diabetes Mellitus (T1DM)
Brief Title: ACZ885 in Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885I2208; 2010-020166-20 (EudraCT Number)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus; Diabetes Type 1
Keywords: ACZ885; diabetes; type 1; C-peptide
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ACZ885 (Experimental)
  Interventions: Drug: ACZ885
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACZ885
  Arms: ACZ885
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of ACZ885 on stimulated C-peptide during a mixed meal test in patients with newly-diagnosed type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes within 3 months of visit 1 and on a stable insulin regimen
* presence of at least one diabetes-related autoantibody
* qualifying C-peptide value in a mixed meal test at visit 1
* willing to not have vaccination with a live vaccine for 18 months, from 3 months before visit 1 until 3 months after the last dose of study drug
* body weight of at least 30 kg

Exclusion Criteria:

* women of child-bearing potential unless a highly effective method of birth control is used (such as combined oral contraceptives, intrauterine devices, etc)
* immunodeficiency
* active infections or febrile illness within 3 days before visit 1
* major dental work within 8 days before visit 1
* positive test for tuberculosis at visit 1
* use of medications other than insulin for the treatment of diabetes Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Measure: Change from baseline of stimulated C-peptide after a mixed meal tolerance test at 13 months | at 13 months

SECONDARY OUTCOMES:
Measure: Change from baseline of stimulated C-peptide after a mixed meal tolerance test at 4, 7, 10, 18, 24, 30 and 36 months | 36 months
Measure: Change from baseline of fasted C-peptide at 4, 7, 10, 13, 18, 24, 30 and 36 months | 36 months
Measure: number of hypoglycemic events | 36 months
Measure: daily insulin dose | 36 months
Measure: anti-ACZ885 antibodies | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Aurora St Luke's Medical Center, Endocrine & Diabetes Center, Milwaukee, Wisconsin, United States
- Canada (2):
  - LMC Endocrinology Centres (Barrie) Ltd, Barrie, Ontario
  - LMC Endocrinology Centres (Bayview) Ltd, Toronto, Ontario
- Germany (3):
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Neuwied
- United Kingdom (4):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Liverpool